CLINICAL TRIAL: NCT05791149
Title: Epigenetic Biomarkers in the Saliva for the Diagnosis of Squamous Cells Carcinoma of the Oral Cavity
Acronym: EPSACO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PI2022_843_0042
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Oral Squamous Cell Carcinoma; Maxillo-facial Surgery; Biomarkers; Saliva; DNA Methylation; Epigenetics
Keywords: Oral Squamous Cell Carcinoma; Maxillo-facial surgery; Biomarkers; Saliva; DNA Methylation; epigenetics
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OSCC patients (Experimental)
  Interventions: Diagnostic Test: saliva tube
- controls (Active Comparator)
  Interventions: Diagnostic Test: saliva tube

INTERVENTIONS:
Diagnostic Test: saliva tube — 1 tube of saliva (~2 ml) will be collected from all patients enrolled in the study. For operated OSCC patients a second tube will be collected during the routine hospital visit 4 weeks after surgery

SUMMARY:
Head and neck squamous cell carcinoma (HNSCC) are malignant tumors originating from the epithelial mucosa of the upper aerodigestive tract. The oral cavity is the most frequent location of HNSCC (oral squamous cell carcinoma: OSCC). Tobacco use and alcohol consumption are the greatest risk factors. The Hauts de France region has one of the highest incidence rates of OSCC. The overall survival of patients with OSCC remains low, with a 5-year overall survival rate of around 60%. In addition to the oncological prognosis, OSCCs and their treatment have a significant impact on the quality of life of patients. An early diagnosis of OSCC is recommended, but it remains difficult. It can be for example challenging to diagnose OSCC in a context of oral premalignant lesions. Identifying objective biomarkers of malignancy would be an advantage and would allow better progress in the field of precision medicine and surgery for these tumors.

The investigators propose to establish the diagnostic use of an optimized DNA methylation profile detected in the saliva of OSCC patients by comparing these epigenetic marks before and after tumor resection.

The investigators will construct a consolidated signature of 4 genes whose DNA is subject to methylation and gene expression is restricted to cancer cells, by crossing TCGA analysis with single-cell analysis (single-cell RNA sequencing).

The investigators propose to analyse DNA methylation of the corresponding genes in the saliva of n=30 OSCC patients recruited for primary surgical resection in the Department of Maxillofacial Surgery vs controls. In addition, the investigators will examine the methylation profiles before / after complete excisional surgery of OSCC. This pilot study will aim to validate the analysis of DNA methylation markers in saliva of OSCC, with the aim of improving the diagnostic precision of OSCC and, secondly, to compare these markers before and after treatment by primary surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient group:
* Patients from the maxillofacial surgery department treated for a histologically confirmed squamous cell carcinoma of the oral cavity
* Patients whose first-line treatment decision at the multidisciplinary meeting in the service of Maxillofacial Surgery is surgery
* Patients who have not yet been treated surgically or by neoadjuvant treatment
* Patients over 18 years old
* Patients who have provided free and informed consent in writing
* Patients benefiting from a social security scheme

Control group:

* Patients in the maxillofacial surgery department not covered for head and neck cancer
* Patients over 18 years old
* Patients who have provided free and informed consent in writing
* Patients benefiting from a social security scheme
* Control group homogeneous with the patient group according to age, sex, tobacco and alcohol consumption

Exclusion Criteria:

* Patients with other types of cancer
* Patients under the age of 18
* Pregnant or breastfeeding women
* Patients under guardianship, curators, legal protection or deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of methylated gene in both groups : control and OSCC patients | one year

SECONDARY OUTCOMES:
Percentage of methylated gene in OSCC patients before surgery | one year
Percentage of methylated gene in OSCC patients after surgery | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Amiens University Hospital, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No